CLINICAL TRIAL: NCT07361016
Title: Comparison of Laparoscopic and Open Total Mesocolic Excision With Central Vascular Ligation for Right Colon Carcinoma
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Mohamed Gohar, assistant lecturer, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: laparoscpic colon cancer
Record Dates: First submitted 2025-12-20; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Right-sided Colon Cancer; Colon Adenocarcinoma; Colorectal Neoplasms
MeSH Terms: conditions — Colonic Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Comparison study
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Open CME with CVL (Active Comparator)
  Interventions: Procedure: open rt hemicolectmy
- Laparoscopic CME with CVL (Active Comparator)
  Interventions: Procedure: right hemicolectomy laparoscopic surgery

INTERVENTIONS:
Procedure: right hemicolectomy laparoscopic surgery — Laparoscopic right hemicolectomy or extended right hemicolectomy using complete mesocolic excision with central vascular ligation, pneumoperitoneum 12-14 mmHg via umbilical port, diamond-shaped port placement, medial-to-lateral dissection along embryological planes, ligation of ileocolic (and right colic/middle colic branch when indicated) at origin, intra- or extracorporeal stapled ileotransverse anastomosis, specimen extraction through Pfannenstiel or right subcostal incision, standard perioperative care.
  Arms: Laparoscopic CME with CVL
Procedure: open rt hemicolectmy — Open right hemicolectomy or extended right hemicolectomy using complete mesocolic excision with central vascular ligation, via midline laparotomy, lateral-to-medial mobilization, ligation of ileocolic (and right colic/middle colic branch when indicated) at origin, extracorporeal ileotransverse anastomosis with hand-sewn sutures, standard perioperative care.
  Arms: Open CME with CVL

SUMMARY:
The goal of this observational comparative study is to assess whether laparoscopic complete mesocolic excision with central vascular ligation (L-CME with CVL) provides improved short-term surgical outcomes compared with open complete mesocolic excision with central vascular ligation (O-CME with CVL) in patients with right-sided colon cancer.

The primary questions this study aims to answer are:

Does laparoscopic CME with CVL reduce blood loss, postoperative complications, and length of hospital stay compared with open CME?

Does laparoscopic CME with CVL achieve equivalent surgical specimen quality and short-term oncological outcomes compared to the open approach?

Researchers compared laparoscopic versus open right hemicolectomy with CME and CVL in adult patients diagnosed with right colon cancer who were eligible for elective surgical resection.

Participants underwent standard preoperative assessment, including clinical evaluation, laboratory testing, imaging studies, colonoscopy, and biopsy confirmation. Surgical treatment consisted of either laparoscopic or open complete mesocolic excision with central vascular ligation, performed according to standardized oncologic surgical principles. Postoperative care followed an enhanced recovery protocol.

Primary outcome measures included operative time, intraoperative blood loss, time to first flatus, postoperative complications, and duration of hospital stay. Secondary outcomes included quality of the surgical specimen (lymph node yield, mesocolic integrity, and margin status) and short-term oncologic outcomes, including early recurrence during follow-up.

ELIGIBILITY:
Inclusion Criteria:

* rt cancer colon

Exclusion Criteria:

* metastatisis

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 22 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Length of Postoperative Hospital Stay | From surgery until discharge (up to 30 days)
  Number of days from the date of surgery to the date of hospital discharge.
Overall Postoperative Morbidity ( Incidence of postoperative complications) | Up to 30 days after surgery
  Occurrence of any postoperative complication, including wound infection, anastomotic leak, abdominal collection, pulmonary infection, urinary tract infection, or deep vein thrombosis, occurring within the early postoperative period.
Intraoperative Blood Loss ( Estimated blood loss (milliliters)) | During surgery
  Volume of blood lost during surgical resection, measured intraoperatively.
Operative Time ( Duration of surgery (minutes)) | During surgery
  Time from skin incision to skin closure.
Postoperative Recovery of Bowel Function (Time to first passage of flatus (hours)) | Up to 72 hours postoperatively
  Time elapsed from completion of surgery to first postoperative flatus, indicating recovery of gastrointestinal motility.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed MM Gohar, Principal Investigator — Kafr Elsheikh university hospitals
Locations (1):
- Kafrelsheikh University, Kafr ash Shaykh, Kafrelsheikh, Egypt

IPD SHARING:
Plan to Share IPD: Yes
comparison study
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 12/12/2022 to 12/12/2024
Access Criteria: anyone

REFERENCES:
- [Background] Hohenberger W, Weber K, Matzel K, Papadopoulos T, Merkel S. Standardized surgery for colonic cancer: complete mesocolic excision and central ligation--technical notes and outcome. Colorectal Dis. 2009 May;11(4):354-64; discussion 364-5. doi: 10.1111/j.1463-1318.2008.01735.x. Epub 2009 Nov 5. PMID 19016817